CLINICAL TRIAL: NCT01453218
Title: Single Centre, Prospective, Open, Non Controlled, Pilot Study for Efficacy and Security Evaluation of Low Nephrotoxicity Immunosuppression, Based on the Use of ATeGe in Liver Transplant Recipients With Pre-transplant Renal Dysfunction
Brief Title: Safety Use of ATeGe in Liver Transplant Recipients With Pre-transplant Renal Dysfunction
Acronym: ATG_HVH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Vall d'Hebron (Other)
Collaborators: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Principal Investigator, Cristina Dopazo Taboada, Consultant and Liver Surgeon, Hospital Vall d'Hebron
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ATG-IRA-HVH.10; 2011-000691-34 (EudraCT Number)
Record Dates: First submitted 2011-10-11; First posted 2011-10-17 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Renal Insufficiency
Keywords: Renal insufficiency; Liver transplant; Acute rejection; Infections; Hepatitis C recurrence
MeSH Terms: conditions — Renal Insufficiency; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Basiliximab (No Intervention): Historical comparable cohort treated with Basiliximab 20mg iv administered at 0 and 4th day post-transplant
- ATeGe-Fresenius (Active Comparator)
  Interventions: Drug: ATeGe-Fresenius

INTERVENTIONS:
Drug: ATeGe-Fresenius — Administered at 1 , 3, 5 and 7 day post-transplant at 2-3mg/kg with dose adjustment according to CD2/CD3 levels
  Arms: ATeGe-Fresenius

SUMMARY:
Renal dysfunction in the context of liver transplantation is a major issue, with difficult patients' management and determining a worsened prognosis.

Physiopathologically pretransplant renal dysfunction is dependent on multifactorial causes, including hypoperfusion-derived functional renal insufficiency, hepatorenal syndrome or interstitial parenchymatous insufficiency. On top, intra- or post-transplant events, including hypoperfusion or calcineurin inhibitors nephrotoxicity may aggravate this situation.

At present MELD criteria favours allocation of organs to patients suffering from renal insufficiency, so at least 30% of the investigators liver transplant patients suffer from some degree of renal impairment pretransplant.

After liver transplant impaired renal function tends to recover partially or completely, unless advanced parenchymatous lesions are significantly involved as a major cause of renal dysfunction.

In this context, calcineurin inhibitors avoiding or sparing protocols may help in the recovery from renal insufficiency, improving long-term prognosis. The use of anti-CD25 antibodies is a good option, but provides a limited antirejection prophylaxis, limiting the use of these antibodies to a reduced cohort of liver transplant patients.

Polyclonal antibodies might provide an advantage in management of liver transplant patients with renal insufficiency, without increasing acute rejection episodes of the allograft efficacy and security evaluation of low nephrotoxicity immunosuppression, based on the use of ATeGe, in liver transplant candidates with pre-transplant renal dysfunction.

The aim of this study is to evaluate the efficacy and security use of immunosuppression based on ATeGe in liver transplant recipients with pre-transplant renal dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate pre-transplant renal dysfunction as defined serum creatinine levels higher than 1.5 mg/dl or eGFR (MDRD-4) <60ml/min.
* First liver transplant, including splits liver transplant.
* Patients aged 18-70 years
* Without a prior contraindication for protocol biopsy of allograft.

Exclusion Criteria:

* Multiorgan transplantation and/or liver transplant from DCD and/or with ABO incompatibility.
* Uncontrolled concomitant infections (including HIV seropositivity) and/or diarrhoea, vomiting or active gastric ulcer.
* Fulminant hepatic insufficiency as first indication for liver transplant
* Hemodynamic instability prior to liver transplant.
* Recipient presenting present or previous neoplasia, except for non-metastatic basal or squamous cutaneous carcinoma or localized hepatocarcinoma with diameter <5 cm or < 3 known lesions with diameter <3 cm.
* Intolerance to study medication.
* Patients having received vaccination with attenuated living vaccines within the previous 4 weeks.
* Severe leukopenia (< 1.2 X 10E9/L) and/or thrombocytopenia (< 50x10E9/L) and/or lymphocyte counts (CD2+/CD3+) less than 10 cells/µl.
* Significant comorbidity.
* Breastfeeding or female patients at fertile age without negative pregnancy test and accepting the use of reliable fertility control method.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Renal function improvement after liver transplant | Measurement will be performed at 1st, 2nd, 3rd, 4th, 5th, 6th, 7th, 14th and 28th day post-transplant, and 2nd, 3rd, 6th and 12th month post-transplant
  Creatinine (mg/dL) and MDRD Glomerular Filtrate Rate (ml/min/1.73m2) will be measured following the time frame described above

SECONDARY OUTCOMES:
Incidence of biopsy proven acute cellular rejection. | Evaluation at 1st , 3rd, 6th, 9th and 12th month post-transplant
  If liver dysfunction is detected, percutaneous liver biopsy will be performed and histological severity will be assed following BANF criteria
Patient and graft survival rates after 12 months, causes of death and retransplant | Evaluation at 1st , 3rd, 6th, 9th and 12th month post-transplant
Relationship between ATeGe doses, immunological variables (lymphocyte counts) and clinical adverse events (acute rejection,infections, HCV recurrence and de novo tumor) | Evaluation at 1st , 3rd, 6th, 9th and 12th month post-transplant
Incidence and severity of HCV infection recurrence, based on clinical and histological criteria. | Once liver dysfunction is detected and one year post-transplant by protocol.
Evaluation of metabolic complications (diabetes mellitus, arterial hypertension and dyslipidemia) | Evaluation at 1st , 3rd, 6th, 9th and 12th month post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: ITXARONE BILBAO, PhD/MD, Principal Investigator — Department of HPB Surgery and Transplants, Hospital Vall d´Hebron (Barcelona, Spain); RAMON CHARCO, PHD/MD, Study Director — Department of HPB Surgery and Transplants, Hospital Vall d´Hebron (Barcelona, Spain); CRISTINA DOPAZO, PhD/MD, Study Chair — Department of HPB Surgery and Transplants, Hospital Vall d´Hebron (Barcelona, Spain); MONICA MARTINEZ, PhD/MD, Study Chair — Department of Inmunology, Hospital Vall d´Hebron (Barcelona, Spain); GONZALO SAPISOCHIN, PhD/MD, Study Chair — Department of HPB Surgery and Transplants, Hospital Vall d´Hebron (Barcelona, Spain); JOSE L LAZARO, MD, Study Chair — Department of HPB Surgery and Transplants, Hospital Vall d´Hebron (Barcelona, Spain); HELENA ALLENDE, PhD/MD, Study Chair — Department of Histology, Hospital Vall d´Hebron (Barcelona, Spain)
Locations (1):
- Department of HPB Surgery and Transplants, Hospital Vall d´Hebron, Barcelona, Spain

REFERENCES:
- [Background] Uemura T, Schaefer E, Hollenbeak CS, Khan A, Kadry Z. Outcome of induction immunosuppression for liver transplantation comparing anti-thymocyte globulin, daclizumab, and corticosteroid. Transpl Int. 2011 Jul;24(7):640-50. doi: 10.1111/j.1432-2277.2011.01250.x. Epub 2011 Mar 23. PMID 21429047
- [Background] Benitez CE, Puig-Pey I, Lopez M, Martinez-Llordella M, Lozano JJ, Bohne F, Londono MC, Garcia-Valdecasas JC, Bruguera M, Navasa M, Rimola A, Sanchez-Fueyo A. ATG-Fresenius treatment and low-dose tacrolimus: results of a randomized controlled trial in liver transplantation. Am J Transplant. 2010 Oct;10(10):2296-304. doi: 10.1111/j.1600-6143.2010.03164.x. PMID 20883560
- [Background] Soliman T, Hetz H, Burghuber C, Gyori G, Silberhumer G, Steininger R, Muhlbacher F, Berlakovich GA. Short-term induction therapy with anti-thymocyte globulin and delayed use of calcineurin inhibitors in orthotopic liver transplantation. Liver Transpl. 2007 Jul;13(7):1039-44. doi: 10.1002/lt.21185. PMID 17600336
- [Background] Soliman T, Hetz H, Burghuber C, Gyori G, Silberhumer G, Steininger R, Muhlbacher F, Berlakovich GA. Short-term versus long-term induction therapy with antithymocyte globulin in orthotopic liver transplantation. Transpl Int. 2007 May;20(5):447-52. doi: 10.1111/j.1432-2277.2007.00463.x. Epub 2007 Mar 2. PMID 17343686
- [Background] Kim MJ, Tsinalis D, Franz S, Binet I, Gurke L, Mihatsch MJ, Steiger J, Thiel G, Dickenmann M. ATG-Fresenius or daclizumab induction therapy in immunologically high risk kidney recipients: a prospective randomized pilot trial. Ann Transplant. 2008;13(4):21-7. PMID 19034219
- [Background] Bajjoka I, Hsaiky L, Brown K, Abouljoud M. Preserving renal function in liver transplant recipients with rabbit anti-thymocyte globulin and delayed initiation of calcineurin inhibitors. Liver Transpl. 2008 Jan;14(1):66-72. doi: 10.1002/lt.21309. PMID 18161842
- [Background] Tector AJ, Fridell JA, Mangus RS, Shah A, Milgrom M, Kwo P, Chalasani N, Yoo H, Rouch D, Liangpunsakul S, Herring S, Lumeng L. Promising early results with immunosuppression using rabbit anti-thymocyte globulin and steroids with delayed introduction of tacrolimus in adult liver transplant recipients. Liver Transpl. 2004 Mar;10(3):404-7. doi: 10.1002/lt.20085. PMID 15004768
- [Derived] Dopazo C, Charco R, Caralt M, Pando E, Lazaro JL, Gomez-Gavara C, Castells L, Bilbao I. Low Total Dose of Anti-Human T-Lymphocyte Globulin (ATG) Guarantees a Good Glomerular Filtration Rate after Liver Transplant in Recipients with Pretransplant Renal Dysfunction. Can J Gastroenterol Hepatol. 2018 Aug 16;2018:1672621. doi: 10.1155/2018/1672621. eCollection 2018. PMID 30186817